CLINICAL TRIAL: NCT03437070
Title: A Phase I Study of Trabectedin in Combination With Fixed Doses of Doxorubicin and Olaratumab in Patients With Metastatic or Recurrent Leiomyosarcoma
Brief Title: Trabectedin, Doxorubicin and Olaratumab in Patients With Metastatic or Recurrent Leiomyosarcoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: University of Miami (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Marilyn Huang, Associate Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170991
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Leiomyosarcoma
Keywords: Advanced Leiomyosarcoma; Recurrent Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Trabectedin; Doxorubicin; olaratumab

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TDO Dose Level (Experimental): Trabectedin [T], Doxorubicin [D], and Olaratumab [O]
  Interventions: Drug: Trabectedin; Drug: Doxorubicin; Drug: Olaratumab

INTERVENTIONS:
Drug: Trabectedin — Administered intravenously per protocol on Day 1 for 21-day cycles.
  Other Names: Yondelis
Drug: Doxorubicin — Administered intravenously per protocol on Day 1 for 21-day cycles.
  Other Names: Doxorubicin Hydrochloride
Drug: Olaratumab — Administered intravenously per protocol
  Other Names: Lartruvo

SUMMARY:
This study seeks to determine if addition of trabectedin (T) to combination doxorubicin (D) and olaratumab (O), is feasible and tolerable with antitumor activity in metastatic or recurrent Leiomyosarcomas (LMS) patients who have limited therapeutic options.

DETAILED DESCRIPTION:
This is a traditional 3+3 phase I trial design to identify the recommended phase II dose (RP2D) of Trabectedin [T] that can be used in combination with Doxorubicin [D] and Olaratumab [O] for the treatment of patients with advanced stage or recurrent LMS.

Patients will be treated at an assigned dose level of combination therapy per dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic, advanced, or recurrent, LMS. Note: Patients should have tissue, either archival or fresh biopsy, submitted for pathologic review to confirm diagnosis of LMS. For patients with recurrent disease with disease free interval greater than six months, a fresh biopsy must be obtained.
2. All patients with recurrent or metastatic LMS deemed unresectable must have measurable disease as defined by RECIST 1.1.

   All patients with advanced LMS may be enrolled after an initial cytoreductive surgery if there is measurable disease as defined by RECIST 1.1.
3. Life expectancy greater than 3 months.
4. Male or female, age ≥18 years
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1.
6. Resolution of clinically significant toxic effects of prior surgery, radiotherapy or systemic anticancer therapy.
7. Patients must not have received prior doxorubicin chemotherapy; only 1 prior chemotherapy line allowable and must be discontinued at least 4 weeks prior to first day of study treatment.
8. Patients should be free of active infections requiring antibiotics (with exception of urinary tract infection).
9. Patients must have adequate organ and marrow function as defined below: Absolute neutrophil count (ANC) ≥1,500 cells/mm³

   * Platelet count ≥100,000/mm³
   * Hemoglobin ≥9.0g/dL
   * Total bilirubin <1.0 upper limit of normal (ULN)
   * Alkaline phosphatase of non-osseous origin ≤ 2.5 x ULN
   * Aminotransferase (AST and ALT) ≤ 2.5 x ULN
   * Creatinine phosphokinase (CPK) ≤ 2.5 x ULN
   * Isotope Dilution Mass Spectrometry (IDMS) creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 40 mL/min
   * Albumin ≤ 3 g/dL*
   * *Hypoalbuminemia < 3 g/dL should be considered carefully but in and of itself, not exclusionary.
10. Women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation until 3 months for women and 5 months for men after completion of study drug administration. WOCBP must have a negative serum or urine test at time of enrollment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study therapy, and 5 months after completion of study drug administration.
11. Patients must have adequate cardiac function (ejection fraction ≥ 45%) to receive therapy.
12. Ability to understand the investigational nature, potential risks and benefits of the research study and to provide valid written informed consent.

Exclusion Criteria:

1. Patients without histologically confirmed LMS
2. Patients without measurable disease by RECIST 1.1 criteria
3. Prior doxorubicin, trabectedin, or olaratumab chemotherapy
4. Patients with an ECOG of 2, 3 or 4 (Appendix C)
5. Patient with known allergies to pegfilgrastim/filgrastim.
6. Patients with known active central nervous system (CNS) metastasis and/or carcinomatous meningitis.
7. Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study therapy and during the study.
8. Patients with a known sensitivity to humanized antibodies or sensitivity attributed to compounds of similar chemical or biological composition to alkylating agents or anthracyclines.
9. A QT interval corrected for heart rate using the Bazett's formula (QTcB) ≥ 480 msec.
10. Patients on combination antiretroviral therapy are ineligible.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infections (including viral hepatitis), decompensated cirrhosis or chronic liver disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
12. Adults unable to consent, pregnant or nursing women or prisoners.
13. Any serious medical or psychiatric illness/condition likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.
14. Diagnosis of another primary malignancy within the past 5 years with the exception of non-melanoma skin cancer.
15. Patients with a prior history of grade 3 capillary leak syndrome (CLS) or <grade 3 CLS with pulmonary involvement.
16. Unwilling to abstain from alcohol ingestion for duration of the study
17. Patients with elevated liver function or bilirubin not meeting criteria for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of Trabectedin in Combination with Doxorubucin and Olaratumab | About 21 days, one cycle of protocol therapy
  Determination of the recommended phase 2 dose (RP2D) of Trabectedin [T] to be used in combination with Doxorubicin [D] and Olaratumab [O] for the treatment of patients with metastatic or recurrent LMS. Patients will be treated at one of 4-6 dose levels according to the standard dose escalation/de-escalation scheme. In accordance with this scheme, the RP2D of TDO will be established as the highest dose level tested for which no more than 2 out of 12 patients experiences dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Toxicity in Study Participants | Up to 8 months
  Determination of the safety, tolerability, and toxicity profile of administering TDO in metastatic or recurrent LMS patients, including assessment of dose-limiting toxicities (DLTs).
Clinical Benefit Rate in Study Participants | From Baseline to End of Treatment, up to 8 months
  Clinical benefit rate (CBR), as defined by best response, (Complete Response (CR), Partial Response (PR) or Stable Disease (SD)) will be assessed using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Huang, MD, MS, Principal Investigator — University of Miami